CLINICAL TRIAL: NCT05707481
Title: Impact of Clinical Pharmacist Led Intervention on Management of Diabetic Hypertensive Patients.
Brief Title: Impact of Clinical Pharmacist-Led Intervention on Management of Diabetic Hypertensive Patients in Eastern Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chettinad Academy of Research and Education (Deemed to be University) (Other)
Collaborators: Purbanchal University (Other)
Responsible Party: Principal Investigator, Dr. Prasanna Dahal, PhD Research Scholar, Chettinad Academy of Research and Education (Deemed to be University)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 382/2022 PhD
Record Dates: First submitted 2023-01-06; First posted 2023-02-01 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Usual Standard Care) (No Intervention): Control group patient will undergo routine care by their physician and nurses. However, the investigator will only provide basic counseling regarding drug prescribed during discharge to the patients. In another term "Usual care" will be provided to the patients
- Intervention Group (Clinical Pharmacist-led educational Intervention) (Other): In addition to routine care by physician and nurses, Patients in interventional group will receive two consecutive face to face interview and counseling of 20-40 minutes during the baseline period and the first follow-up period at 3-month by clinical pharmacist. Teaching and counseling session involves information on various non-pharmacological and pharmacological disease management strategies.
  Interventions: Other: Clinical Pharmacist-Led Educational Intervention

INTERVENTIONS:
Other: Clinical Pharmacist-Led Educational Intervention — Non Pharmacological management strategies include information related to life style modification, healthy dietary habits, physical activity and stress management techniques. In contrast, pharmacological educational intervention involves disease -related information ( diabetes/hypertension sign and symptoms, risk factor, complications, self-monitoring of blood pressure/glucose, symptoms and management of hypoglycemia/hypotension etc. ) and drug related information ( prescribed drug name, indication, contraindication, adverse effects etc.) as well as importance of adherence to prescribed medication and strategies to minimize DRPs issues. These teaching sessions will be carried out with the help of verbal communication, audio visual demonstration (including charts,pictorial etc) and information leaflets. Furthermore, a copy of educational package would be given to each participant for reference and guidance.
  Arms: Intervention Group (Clinical Pharmacist-led educational Intervention)

SUMMARY:
Diabetic-Hypertensives are at a higher risk of premature microvascular and macrovascular complications than diabetes alone. Proper lifestyle management, diet, disease monitoring, and medication adherence is essential in achieving desired therapeutic outcomes, preventing complications and improving those patients' Health-Related Quality of Life (HRQoL). Pharmacists are the most accessible healthcare professionals to the public and have a crucial role in optimizing treatment outcomes in patients with chronic diseases such as diabetes and hypertension. Experimental trials' demonstrating the potential roles of pharmaceutical services is scarce in the literature, particularly in developing countries of south Asia. Therefore, the investigators plan to conduct a prospective-interventional trial to determine the potential impacts of pharmacist-supervised educational intervention on the management of "Type II diabetic with comorbid hypertension" patients. Patient data will be collected using patient's clinical profile forms, General Medication adherence Scale (GMAS), Patients Satisfaction towards pharmaceutical services (PSPSQ), Health Related-KAP questionnaires. Data will be verified, stored, entered into databases, and analyzed according to the data management plan. The findings will be compared in terms of clinical and nonclinical outcome measures between the control and test groups to ascertain the conclusion.

DETAILED DESCRIPTION:
Diabetics are twice as likely as non-diabetics to develop hypertension. Hypertension is a strong predictor of adverse cerebulo-vascular and cardiovascular events in people with diabetes, which increases risk of Premature micro-vascular and macro-vascular problems in patients encompassing both diseases. Therefore, strict glycemic and blood pressure control is essential to subdue complication and prevent dreadful cardiovascular events such as stroke, Ischemia and myocardial infarction. Participants with both chronic diseases may have lower HRQoL due to increased susceptibility towards cardiovascular comorbidities. Adherence to medication is equally crucial for treatment success. Pharmacist in collaboration with other healthcare members, could play a vital role in the care of patients and optimizing treatment outcomes in patients with chronic diseases .

Chronic disease management is of particular interest to clinical pharmacist since most intervention requires long-term prescription medication use. The international pharmaceutical federation (FIP) and world health organization (WHO) have implored pharmacists to support people with chronic disease through their expanded role that includes "pharmaceutical care." In Nepal, Clinical Pharmacy practice is still in early infancy, though few studies have shown encouraging impacts of pharmaceutical care services. Similarly, there is a significant gap in the literature in this region addressing the impact of pharmacist-supervised educational intervention on both clinical and nonclinical outcomes measures, primarily focusing on co-morbid Diabetes- Hypertensive patients. Therefore, these studies are intended to recap and fill that gap area and add new and valuable insight to the available literature.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 40 to 68 years.
* Clinically diagnosed with type II diabetes mellitus with hypertension as co-morbidity.
* Minimum one year of the medical history of diabetic and hypertension.
* Minimum 6 months on antidiabetic as well as antihypertensive medication therapy.
* Patients willing to participate in the study and those providing written informed consent for participation.

Exclusion Criteria:

* Patients with Type I diabetes mellitus, Diabetic insipidus, Gestational diabetes or other forms of diabetes.
* Presence of other chronic disease co-morbidity other than hypertension and diabetes complications.
* Mentally incompetent patients, Pregnant, critically ill patients (requiring hospital admission).
* Patients have tuberculosis, Corona virus, and other highly communicable diseases.
* Those patients not willing to performing routine follow-up visit.

Ages: 40 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-07-04 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | baseline, follow up at 3 months and 6 months respectively
  Assessed with measurement of Systolic and diastolic blood pressure in mmHg using sphygmomanometer
Change in blood glycemic profile | baseline, follow up at 3 months and 6 months respectively
  Assessed with measurement of Fasting Blood Sugar (FBS) and Post Prandial Blood Sugar (PPBS) in mg/dl.
change in glycosylated hemoglobin (HbA1C) level | baseline, follow up at 3 months and 6 months respectively
  assessed from patients glycosylated hemoglobin (HbA1C) level test, measured in percent (%)
Impact of Intervention in Patients Medication Adherence | baseline, follow up at 3 months and 6 months respectively
  It will be measured using translated and validated Nepalese version of the 11-item Novel general medication adherence Scale (GMAS) questionnaire divided into three categories based on a four-level Likert scale. GMAS tools provide a wide range of components, including disease and medication burden, patient behavior both intentional and unintentional, and cost-related burden associated with non-adherence. Higher Scores better the outcomes, measured within categories and overall adherence level.
Compare patients perceived Satisfaction of pharmaceutical care services | baseline, follow up at 3 months and 6 months respectively
  This will be assessed by using Nepali version of Patients Perceived satisfaction of Pharmacist care (PSPSQ. 2 ) questionnaire. This tool comprises 20 items questionnaire divided into three dimensions based on a four-point Likert scale. Dimensions include quality of care, pharmacist-patient relationships, and overall satisfaction. Higher scores represent better outcomes, measured within domains and overall satisfaction levels.
Change in Health related Quality of Life | baseline, follow up at 3 months and 6 months respectively
  Translated Nepali version of Euro 5 D 5 L questionnaire measures will be used to measure patients' health-related quality of life (HRQoL). This questionnaire created by the European Quality of Life Group (EuroQol Group) measure HRQoL in five dimension Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has five levels to describe the severity: no problem, slight problem, moderate problem, severe problem, and unable (very severe). The outcomes will be measured in the overall health utility index value. The index value ranges from -1 to 1 (0 indicates death, <0 indicates worse than death, and 1 indicates full health)

SECONDARY OUTCOMES:
Change in routine clinical laboratory parameters of patients Lipid Profile test. | baseline, follow up at 3 months and 6 months respectively
  Data will be obtained from routine clinical laboratory test of patients blood Lipid Profile ( Total cholesterol, High density lipoprotein (HDL) Cholesterol, Low density lipoprotein (LDL) cholesterol, Very low density lipoprotein (VLDL) Cholesterol, and Triglycerides) measured in mg/dl.
Change in Patients health related Knowledge, Attitude and Practice | baseline, follow up at 3 months and 6 months respectively
  Patient knowledge, attitude and practice will be assessed using 25-item Disease related Health Knowledge, attitude and practice questionnaires developed by Investigators through literature review and content validated with a team of health care professionals. The higher the scores within domains better the outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Prasanna Dahal, PharmD, Principal Investigator — Chettinad Academy of Research and Education (Deemed to be University)
Locations (1):
- Purbanchal University Hospital, Gothgaun,Sundar Haraicha Municipality, Morang, Koshi, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Naqvi AA, Hassali MA, Jahangir A, Nadir MN, Kachela B. Translation and validation of the English version of the general medication adherence scale (GMAS) in patients with chronic illnesses. J Drug Assess. 2019 Feb 6;8(1):36-42. doi: 10.1080/21556660.2019.1579729. eCollection 2019. PMID 30863660
- [Background] Shrestha R, Sapkota B, Khatiwada AP, Shrestha S, Khanal S, Kc B, Paudyal V. Translation, Cultural Adaptation and Validation of General Medication Adherence Scale (GMAS) into the Nepalese Language. Patient Prefer Adherence. 2021 Aug 27;15:1873-1885. doi: 10.2147/PPA.S320866. eCollection 2021. PMID 34475753
- [Background] Sakharkar P, Bounthavong M, Hirsch JD, Morello CM, Chen TC, Law AV. Development and validation of PSPSQ 2.0 measuring patient satisfaction with pharmacist services. Res Social Adm Pharm. 2015 Jul-Aug;11(4):487-98. doi: 10.1016/j.sapharm.2014.10.006. Epub 2014 Oct 22. PMID 25481330
- [Background] Shrestha S, Sapkota B, Thapa S, K C B, Khanal S. Translation, cross-cultural adaptation and validation of Patient Satisfaction with Pharmacist Services Questionnaire (PSPSQ 2.0) into the Nepalese version in a community settings. PLoS One. 2020 Oct 9;15(10):e0240488. doi: 10.1371/journal.pone.0240488. eCollection 2020. PMID 33035243